CLINICAL TRIAL: NCT03175757
Title: A Randomized, Single-blind, Placebo-controlled Study to Evaluate the Effects of a Turmeric and Black Cumin Seed Formulation on Cholesterol Levels Among Generally Healthy Participants
Brief Title: A Study to Evaluate the Effects of a Turmeric and Black Cumin Seed Formulation on Cholesterol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CL086
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Cholesterol Health
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholesterol Health Formulation (Experimental): Turmeric and black cumin seed preparation
  Interventions: Dietary Supplement: Turmeric and Black Cumin Seed
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmeric and Black Cumin Seed — Turmeric and Black Cumin Seed formulation
  Arms: Cholesterol Health Formulation
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of a turmeric and black cumin seed formulation on cholesterol levels.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, placebo-controlled study to evaluate the effects of a turmeric and black cumin seed formulation on cholesterol levels. Each subject will receive a specific dose of the formulation or placebo twice daily. Participants will undergo assessments of blood tests, vital signs, body weight, waist circumference, hip circumference and waist-to-hip ratio with completion of a questionnaire.

The primary objective of the study is to assess the effects of the turmeric and black cumin seed formulation on fasting levels of Total Cholesterol.

Secondary objectives include assessment of the effects of turmeric and black cumin seed formulation on: fasting levels of: LDL Cholesterol, parameters in the NMR LipoProfile®, Oxidized LDL, Triglycerides, HDL cholesterol, C-reactive protein, blood glucose, Insulin and Hemoglobin A1c, as well as the assessments of the values/scores of body weight, waist circumference, hip circumference, waist-to-hip ratio, blood pressure and the SF-36 survey scores.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, between 40 and 75 years of age
2. Meeting one of the following two criteria:

   1. Having a BMI between 25.0 and 34.9
   2. Waist circumference > 40.0 inches in males and > 35.0 inches in females
3. Having Total Cholesterol levels at Baseline/screening of between 190 and 239 mg/dl
4. Generally healthy and having no difficulty with digestion or absorption of food
5. Willing and able to give written informed consent
6. Clearly understands the procedures and requirements for the study
7. Able to maintain stable physical activity and dietary habits throughout the study
8. Willing and able to comply with all study procedures and data recording obligations
9. Having the capability of communicating, including reading in English

Exclusion Criteria:

1. Having smoked any cigarette, electronic cigarette, cigar, pipe, or recreational drug in the past 30 days
2. History of allergy or sensitivity to any component of the study products
3. Donation of blood within 30 days prior Baseline/screening
4. Participation in another study within 30 days prior to Baseline/screening
5. Being pregnant, planning on becoming pregnant during study participation or breast feeding
6. Having the following medical condition(s): diabetes, hypotension, hypertension (changed antihypertensive medication or dose in the preceding 3 months and/or likely to do so during the study), cardiovascular disease (arrhythmia, edema with or without congestive heart failure, heart attack, stroke, abnormal EKG), gastrointestinal disease requiring daily prescribed medication (gastroesophageal reflux, gastritis, and peptic or duodenal ulcer), gallbladder disease or gallstones, biliary obstruction (past or present), endocrine disease (hyper- or hypothyroidism), psychiatric disorder (anxiety if untreated, eating disorder) neurologic disease (Parkinson's disease, intracranial hemorrhage, head injury, brain tumor, evidence of delirium, confusion, dementia, Alzheimer's disease, migraine headache (if last migraine headache was < 3 years prior to Baseline/screening), urologic disease, chronic inflammatory or autoimmune disease, cancer (unless skin cancer other than melanoma which has been treated > 3 years prior to Baseline/screening), liver and kidney disease, insomnia, blood coagulation disorder (anemia, thrombus, embolism), sleep apnea, or other condition(s) that would preclude participation in the study in the judgment of the investigator/sub-investigator (Sub-I).
7. Currently taking or having taken cholesterol-lowering medication(s) including HMGCR inhibitors, cholesterol binding resins, fibrates, or nicotinic acid >1 gram/day within 30 days prior to screening
8. Currently taking or having taken a supplemental product that may affect cholesterol levels (red yeast rice, red mold dioscorea, guggulipid, policosanol, pantethine, beta-sitosterol, artichoke leaf, or supplemental fiber) within 30 days prior to Baseline/screening
9. Currently taking or having taken a fish oil or krill oil product within 30 days prior to Baseline/screening
10. Currently taking or having taken anxiolytics and sedative hypnotics, anticonvulsants, antineoplastics, anti-migraine medication(s), opioid analgesics, monoamine oxidase inhibitors (MAOIs), phosphodiesterase inhibitors, adenosine reuptake inhibitors, dopamine agonists, dopamine antagonists, or immunosuppressants within 30 days prior to Baseline/screening
11. Currently talking or having taken anti-inflammatory medication(s) within 14 days prior to screening (unless on a stable daily dose of aspirin 81mg for 3 months prior to screening and not likely to change dose during the study) or in the judgment of the PI/Sub-I would not preclude participation in the study
12. Having had a surgical procedure, pacemaker or any internal medical device other than artificial joints which, in the judgment of the PI/Sub-I, would preclude participation in the study
13. Having had a routine dental cleaning or other dental procedure within 14 days prior to Baseline/screening
14. Having screening laboratory test values: bilirubin > 2.5 x ULN, AST/SGOT and ALT/SGPT > 2.5 x ULN, serum creatinine > 1.5 mg/dL, blood glucose > 125 mg/dL, or any other lab test result(s) that would preclude participation in the study in the judgment of the PI/Sub-I
15. Having blood pressure readings at Baseline/screening > 140 systolic or > 90 diastolic on two consecutive readings unless permitted to proceed to the next visit in the judgment of the PI/Sub-I
16. Currently consumes more than 6 standard alcoholic drinks per week (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
17. History of known alcohol or substance abuse (e.g., opiates, benzodiazepines, or amphetamines)
18. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges and tangelos
19. Having any other significant circumstance that would preclude study participation in the judgment of the PI/Sub-I

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | 60 days
  Mean change from Baseline/screening to Day 60

SECONDARY OUTCOMES:
LDL Cholesterol | 60 days
  Mean change from Baseline/screening to Day 60
Oxidized LDL | 60 days
  Mean change from Baseline/screening to Day 60
Triglycerides | 60 days
  Mean change from Baseline/screening to Day 60
HDL Cholesterol | 60 days
  Mean change from Baseline/screening to Day 60
C-reactive protein (hs-CRP) | 60 days
  Mean change from Baseline/screening to Day 60
Blood glucose | 60 days
  Mean change from Baseline/screening to Day 60
Insulin | 60 days
  Mean change from Baseline/screening to Day 60
Hemoglobin A1C | 60 days
  Mean change from Baseline/screening to Day 60
Body weight | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
Blood pressure | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
SF-36 health survey scores | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
Waist circumference | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
Hip circumference | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
Waist-to-Hip ratio | 60 days
  Mean change from Day 1 (Enrollment) to Day 60
LDL-P (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
LDL-C (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
HDL-C (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
Triglycerides (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
Cholesterol, Total (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
HDL-P (Total) (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
Small LDL-P (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
LDL Size (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60
LP-IR Score (NMR Lipoprofile) | 60 days
  Mean change from Baseline/screening to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joyal, M.D., Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad S, Beg ZH. Hypolipidemic and antioxidant activities of thymoquinone and limonene in atherogenic suspension fed rats. Food Chem. 2013 Jun 1;138(2-3):1116-24. doi: 10.1016/j.foodchem.2012.11.109. Epub 2012 Dec 5. PMID 23411222
- [Background] Al-Naqeep G, Al-Zubairi AS, Ismail M, Amom ZH, Esa NM. Antiatherogenic Potential of Nigella sativa Seeds and Oil in Diet-Induced Hypercholesterolemia in Rabbits. Evid Based Complement Alternat Med. 2011;2011:213628. doi: 10.1093/ecam/neq071. Epub 2011 Jun 16. PMID 21792359
- [Background] Ali BH, Blunden G. Pharmacological and toxicological properties of Nigella sativa. Phytother Res. 2003 Apr;17(4):299-305. doi: 10.1002/ptr.1309. PMID 12722128
- [Background] Amin F, Gilani AH, Mehmood MH, Siddiqui BS, Khatoon N. Coadministration of black seeds and turmeric shows enhanced efficacy in preventing metabolic syndrome in fructose-fed rats. J Cardiovasc Pharmacol. 2015 Feb;65(2):176-83. doi: 10.1097/FJC.0000000000000179. PMID 25384193
- [Background] Amin F, Islam N, Anila N, Gilani AH. Clinical efficacy of the co-administration of Turmeric and Black seeds (Kalongi) in metabolic syndrome - a double blind randomized controlled trial - TAK-MetS trial. Complement Ther Med. 2015 Apr;23(2):165-74. doi: 10.1016/j.ctim.2015.01.008. Epub 2015 Jan 14. PMID 25847554
- [Background] Asgary S, Sahebkar A, Goli-Malekabadi N. Ameliorative effects of Nigella sativa on dyslipidemia. J Endocrinol Invest. 2015 Oct;38(10):1039-46. doi: 10.1007/s40618-015-0337-0. Epub 2015 Jul 2. PMID 26134064
- [Background] Bamosa AO, Ali BA, al-Hawsawi ZA. The effect of thymoquinone on blood lipids in rats. Indian J Physiol Pharmacol. 2002 Apr;46(2):195-201. PMID 12500494
- [Background] Carroll RE, Benya RV, Turgeon DK, Vareed S, Neuman M, Rodriguez L, Kakarala M, Carpenter PM, McLaren C, Meyskens FL Jr, Brenner DE. Phase IIa clinical trial of curcumin for the prevention of colorectal neoplasia. Cancer Prev Res (Phila). 2011 Mar;4(3):354-64. doi: 10.1158/1940-6207.CAPR-10-0098. PMID 21372035
- [Background] Chen FY, Zhou J, Guo N, Ma WG, Huang X, Wang H, Yuan ZY. Curcumin retunes cholesterol transport homeostasis and inflammation response in M1 macrophage to prevent atherosclerosis. Biochem Biophys Res Commun. 2015 Nov 27;467(4):872-8. doi: 10.1016/j.bbrc.2015.10.051. Epub 2015 Oct 19. PMID 26471308
- [Background] Cheng AL, Hsu CH, Lin JK, Hsu MM, Ho YF, Shen TS, Ko JY, Lin JT, Lin BR, Ming-Shiang W, Yu HS, Jee SH, Chen GS, Chen TM, Chen CA, Lai MK, Pu YS, Pan MH, Wang YJ, Tsai CC, Hsieh CY. Phase I clinical trial of curcumin, a chemopreventive agent, in patients with high-risk or pre-malignant lesions. Anticancer Res. 2001 Jul-Aug;21(4B):2895-900. PMID 11712783
- [Background] Dahri AH, Chandiol AM, Rahoo AA, Memon RA. Effect of Nigella sativa (kalonji) on serum cholesterol of albino rats. J Ayub Med Coll Abbottabad. 2005 Apr-Jun;17(2):72-4. PMID 16092657
- [Background] Dollah MA, Parhizkar S, Latiff LA, Bin Hassan MH. Toxicity effect of nigella sativa on the liver function of rats. Adv Pharm Bull. 2013;3(1):97-102. doi: 10.5681/apb.2013.016. Epub 2013 Feb 7. PMID 24312819
- [Background] Dong SZ, Zhao SP, Wu ZH, Yang J, Xie XZ, Yu BL, Nie S. Curcumin promotes cholesterol efflux from adipocytes related to PPARgamma-LXRalpha-ABCA1 passway. Mol Cell Biochem. 2011 Dec;358(1-2):281-5. doi: 10.1007/s11010-011-0978-z. Epub 2011 Jul 12. PMID 21748336
- [Background] Fan C, Wo X, Dou X, Xu L, Qian Y, Luo Y, Yan J. Regulation of LDL receptor expression by the effect of curcumin on sterol regulatory element pathway. Pharmacol Rep. 2006 Jul-Aug;58(4):577-81. PMID 16963807
- [Background] Haas MJ, Onstead-Haas LM, Naem E, Wong NC, Mooradian AD. Induction of apolipoprotein A-I gene expression by black seed (Nigella sativa) extracts. Pharm Biol. 2014 Sep;52(9):1119-27. doi: 10.3109/13880209.2013.879187. Epub 2014 Mar 17. PMID 24635344
- [Background] Heshmati J, Namazi N. Effects of black seed (Nigella sativa) on metabolic parameters in diabetes mellitus: a systematic review. Complement Ther Med. 2015 Apr;23(2):275-82. doi: 10.1016/j.ctim.2015.01.013. Epub 2015 Feb 9. PMID 25847566
- [Background] Hosseinzadeh H, Parvardeh S, Asl MN, Sadeghnia HR, Ziaee T. Effect of thymoquinone and Nigella sativa seeds oil on lipid peroxidation level during global cerebral ischemia-reperfusion injury in rat hippocampus. Phytomedicine. 2007 Sep;14(9):621-7. doi: 10.1016/j.phymed.2006.12.005. Epub 2007 Feb 8. PMID 17291733
- [Background] Ibrahim RM, Hamdan NS, Ismail M, Saini SM, Abd Rashid SN, Abd Latiff L, Mahmud R. Protective Effects of Nigella sativa on Metabolic Syndrome in Menopausal Women. Adv Pharm Bull. 2014;4(1):29-33. doi: 10.5681/apb.2014.005. Epub 2013 Dec 23. PMID 24409406
- [Background] Kaatabi H, Bamosa AO, Lebda FM, Al Elq AH, Al-Sultan AI. Favorable impact of Nigella sativa seeds on lipid profile in type 2 diabetic patients. J Family Community Med. 2012 Sep;19(3):155-61. doi: 10.4103/2230-8229.102311. PMID 23230380
- [Background] Kuptniratsaikul V, Dajpratham P, Taechaarpornkul W, Buntragulpoontawee M, Lukkanapichonchut P, Chootip C, Saengsuwan J, Tantayakom K, Laongpech S. Efficacy and safety of Curcuma domestica extracts compared with ibuprofen in patients with knee osteoarthritis: a multicenter study. Clin Interv Aging. 2014 Mar 20;9:451-8. doi: 10.2147/CIA.S58535. eCollection 2014. PMID 24672232
- [Background] Lin XL, Liu MH, Hu HJ, Feng HR, Fan XJ, Zou WW, Pan YQ, Hu XM, Wang Z. Curcumin enhanced cholesterol efflux by upregulating ABCA1 expression through AMPK-SIRT1-LXRalpha signaling in THP-1 macrophage-derived foam cells. DNA Cell Biol. 2015 Sep;34(9):561-72. doi: 10.1089/dna.2015.2866. Epub 2015 Jun 23. PMID 26102194
- [Background] Liu T, Li C, Sun H, Luo T, Tan Y, Tian D, Guo Z. Curcumin inhibits monocyte chemoattractant protein-1 expression and enhances cholesterol efflux by suppressing the c-Jun N-terminal kinase pathway in macrophage. Inflamm Res. 2014 Oct;63(10):841-50. doi: 10.1007/s00011-014-0758-9. Epub 2014 Jul 27. PMID 25064633
- [Background] Mirzabeigi P, Mohammadpour AH, Salarifar M, Gholami K, Mojtahedzadeh M, Javadi MR. The Effect of Curcumin on some of Traditional and Non-traditional Cardiovascular Risk Factors: A Pilot Randomized, Double-blind, Placebo-controlled Trial. Iran J Pharm Res. 2015 Spring;14(2):479-86. PMID 25901155
- [Background] Mooradian AD, Haas MJ. The effect of nutritional supplements on serum high-density lipoprotein cholesterol and apolipoprotein A-I. Am J Cardiovasc Drugs. 2014 Aug;14(4):253-74. doi: 10.1007/s40256-014-0068-1. PMID 24604774
- [Background] Morrone Mda S, Schnorr CE, Behr GA, Gasparotto J, Bortolin RC, da Boit Martinello K, Saldanha Henkin B, Rabello TK, Zanotto-Filho A, Gelain DP, Moreira JC. Curcumin Supplementation Decreases Intestinal Adiposity Accumulation, Serum Cholesterol Alterations, and Oxidative Stress in Ovariectomized Rats. Oxid Med Cell Longev. 2016;2016:5719291. doi: 10.1155/2016/5719291. Epub 2015 Nov 23. PMID 26640615
- [Background] Panahi Y, Hosseini MS, Khalili N, Naimi E, Soflaei SS, Majeed M, Sahebkar A. Effects of supplementation with curcumin on serum adipokine concentrations: A randomized controlled trial. Nutrition. 2016 Oct;32(10):1116-22. doi: 10.1016/j.nut.2016.03.018. Epub 2016 Mar 31. PMID 27297718
- [Background] Panahi Y, Kianpour P, Mohtashami R, Jafari R, Simental-Mendia LE, Sahebkar A. Curcumin Lowers Serum Lipids and Uric Acid in Subjects With Nonalcoholic Fatty Liver Disease: A Randomized Controlled Trial. J Cardiovasc Pharmacol. 2016 Sep;68(3):223-9. doi: 10.1097/FJC.0000000000000406. PMID 27124606
- [Background] Peschel D, Koerting R, Nass N. Curcumin induces changes in expression of genes involved in cholesterol homeostasis. J Nutr Biochem. 2007 Feb;18(2):113-9. doi: 10.1016/j.jnutbio.2006.03.007. Epub 2006 May 18. PMID 16713233
- [Background] Ragheb A, Elbarbry F, Prasad K, Mohamed A, Ahmed MS, Shoker A. Attenuation of the development of hypercholesterolemic atherosclerosis by thymoquinone. Int J Angiol. 2008 Winter;17(4):186-92. doi: 10.1055/s-0031-1278307. PMID 22477447
- [Background] Sanmukhani J, Satodia V, Trivedi J, Patel T, Tiwari D, Panchal B, Goel A, Tripathi CB. Efficacy and safety of curcumin in major depressive disorder: a randomized controlled trial. Phytother Res. 2014 Apr;28(4):579-85. doi: 10.1002/ptr.5025. Epub 2013 Jul 6. PMID 23832433
- [Background] Sahebkar A, Beccuti G, Simental-Mendia LE, Nobili V, Bo S. Nigella sativa (black seed) effects on plasma lipid concentrations in humans: A systematic review and meta-analysis of randomized placebo-controlled trials. Pharmacol Res. 2016 Apr;106:37-50. doi: 10.1016/j.phrs.2016.02.008. Epub 2016 Feb 10. PMID 26875640
- [Background] Shafiq H, Ahmad A, Masud T, Kaleem M. Cardio-protective and anti-cancer therapeutic potential of Nigella sativa. Iran J Basic Med Sci. 2014 Dec;17(12):967-79. PMID 25859300
- [Background] Sharma RA, McLelland HR, Hill KA, Ireson CR, Euden SA, Manson MM, Pirmohamed M, Marnett LJ, Gescher AJ, Steward WP. Pharmacodynamic and pharmacokinetic study of oral Curcuma extract in patients with colorectal cancer. Clin Cancer Res. 2001 Jul;7(7):1894-900. PMID 11448902
- [Background] Shuid AN, Mohamed N, Mohamed IN, Othman F, Suhaimi F, Mohd Ramli ES, Muhammad N, Soelaiman IN. Nigella sativa: A Potential Antiosteoporotic Agent. Evid Based Complement Alternat Med. 2012;2012:696230. doi: 10.1155/2012/696230. Epub 2012 Sep 3. PMID 22973403
- [Background] Singh V, Jain M, Misra A, Khanna V, Rana M, Prakash P, Malasoni R, Dwivedi AK, Dikshit M, Barthwal MK. Curcuma oil ameliorates hyperlipidaemia and associated deleterious effects in golden Syrian hamsters. Br J Nutr. 2013 Aug 28;110(3):437-46. doi: 10.1017/S0007114512005363. Epub 2013 May 15. PMID 23673139
- [Background] Singh V, Rana M, Jain M, Singh N, Naqvi A, Malasoni R, Dwivedi AK, Dikshit M, Barthwal MK. Curcuma oil attenuates accelerated atherosclerosis and macrophage foam-cell formation by modulating genes involved in plaque stability, lipid homeostasis and inflammation. Br J Nutr. 2015 Jan 14;113(1):100-13. doi: 10.1017/S0007114514003195. Epub 2014 Nov 13. PMID 25391643
- [Background] Tai MH, Chen PK, Chen PY, Wu MJ, Ho CT, Yen JH. Curcumin enhances cell-surface LDLR level and promotes LDL uptake through downregulation of PCSK9 gene expression in HepG2 cells. Mol Nutr Food Res. 2014 Nov;58(11):2133-45. doi: 10.1002/mnfr.201400366. Epub 2014 Sep 19. PMID 25164566
- [Background] Yang YS, Su YF, Yang HW, Lee YH, Chou JI, Ueng KC. Lipid-lowering effects of curcumin in patients with metabolic syndrome: a randomized, double-blind, placebo-controlled trial. Phytother Res. 2014 Dec;28(12):1770-7. doi: 10.1002/ptr.5197. Epub 2014 Aug 6. PMID 25131839
- [Background] Zaoui A, Cherrah Y, Alaoui K, Mahassine N, Amarouch H, Hassar M. Effects of Nigella sativa fixed oil on blood homeostasis in rat. J Ethnopharmacol. 2002 Jan;79(1):23-6. doi: 10.1016/s0378-8741(01)00342-7. PMID 11744291
- [Background] Zhao JF, Ching LC, Huang YC, Chen CY, Chiang AN, Kou YR, Shyue SK, Lee TS. Molecular mechanism of curcumin on the suppression of cholesterol accumulation in macrophage foam cells and atherosclerosis. Mol Nutr Food Res. 2012 May;56(5):691-701. doi: 10.1002/mnfr.201100735. PMID 22648616
- [Background] Zingg JM, Hasan ST, Meydani M. Molecular mechanisms of hypolipidemic effects of curcumin. Biofactors. 2013 Jan-Feb;39(1):101-21. doi: 10.1002/biof.1072. Epub 2013 Jan 22. PMID 23339042